CLINICAL TRIAL: NCT02401737
Title: A Phase 1b Dose-Ranging Study to Assess the Safety, Pharmacokinetics and Initial Antiviral Efficacy of NVR 3-778 in Patients With HBeAg-Positive Chronic Hepatitis B Virus Infection
Brief Title: Dose-Ranging Study to Assess the Safety, PK and Initial Antiviral Efficacy of NVR 3-778 in Chronic HBV Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novira Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: NVR3-778-101B
Record Dates: First submitted 2015-03-11; First posted 2015-03-30 (Estimated); Last update posted 2017-10-18 (Actual); Status verified 2017-10

CONDITIONS: Chronic Hepatitis B
Keywords: Hepatitis B
MeSH Terms: conditions — Hepatitis B, Chronic; Hepatitis B | interventions — NVR 3-778; peginterferon alfa-2a

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- NVR 3-778 (Experimental): NVR 3-778 in varying doses of capsules by mouth for 28 days
  Interventions: Drug: NVR 3-778
- Placebo for NVR 3-778 (Placebo Comparator): Placebo for NVR 3-778 in varying doses of capsules by mouth for 28 days
  Interventions: Drug: Placebo for NVR 3-778
- NVR 3-778 and Pegasys (Experimental): NVR 3-778 and Pegasys in combination in a yet to be determined dose by mouth and subcutaneous injection for 28 days
  Interventions: Drug: NVR 3-778; Drug: Pegasys
- Pegasys (Active Comparator): Pegasys alone in a yet to be determined dose by subcutaneous injection for 28 days
  Interventions: Drug: Pegasys

INTERVENTIONS:
Drug: NVR 3-778
  Arms: NVR 3-778; NVR 3-778 and Pegasys
Drug: Placebo for NVR 3-778 — Sugar pill manufactured to mimic the NVR 3-778 capsule
  Arms: Placebo for NVR 3-778
Drug: Pegasys
  Other Names: peginterferon alfa-2a
  Arms: NVR 3-778 and Pegasys; Pegasys

SUMMARY:
This Phase 1b trial will assess the dose-related safety and PK profile of different doses of NVR 3-778 in patients with chronic hepatitis B. Additionally,changes in patients' serum HBV DNA levels and other virologic efficacy parameters will be assessed.

DETAILED DESCRIPTION:
The Phase 1b assessments of the dose-related safety, PK, and initial antiviral efficacy of NVR 3-778 in hepatitis B patients will also be conducted at approximately 14 different sites to meet enrollment goals of 54-84 chronic hepatitis B patients.

To promote objective safety and tolerance assessments during this trial, study subjects, and site personnel administering the study drug and performing the clinical assessments on the subjects, will be blinded to individual subjects' treatments assignments (active NVR 3-778 or placebo doses), for all treatment cohorts in the study. Study advancement to subsequent patient cohorts will require satisfactory interim reviews of available cumulative safety data by the Safety Review Committees (SRC), using the safety criteria and review procedures described in the protocol. Also, there will be one interim review of safety data by an independent Safety Monitoring Board (SMB), as described in the protocol.

ELIGIBILITY:
Patients may be male or female between 18 and 65 years of age, with a BMI of 18-35kg/m2. Patients must be HBeAg positive and have chronic hepatitis B with no history of clinical decompensation.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2015-01-31 (Actual); Primary Completion 2016-05-18 (Actual); Study Completion 2016-05-18 (Actual)

PRIMARY OUTCOMES:
Compared with baseline, decline of serum HBV-DNA in the value | Up to 28 days

CONTACTS AND LOCATIONS:
Locations (10):
- United States (4):
  - Costa Mesa, California
  - Pasadena, California
  - San Diego, California
  - San Francisco, California
- Hong Kong, China
- Singapore, Singapore
- South Korea (2):
  - Chuncheon
  - Seongnam
- Taiwan (2):
  - Kaohsiung City
  - Keelung

REFERENCES:
- [Derived] Yuen MF, Gane EJ, Kim DJ, Weilert F, Yuen Chan HL, Lalezari J, Hwang SG, Nguyen T, Flores O, Hartman G, Liaw S, Lenz O, Kakuda TN, Talloen W, Schwabe C, Klumpp K, Brown N. Antiviral Activity, Safety, and Pharmacokinetics of Capsid Assembly Modulator NVR 3-778 in Patients with Chronic HBV Infection. Gastroenterology. 2019 Apr;156(5):1392-1403.e7. doi: 10.1053/j.gastro.2018.12.023. Epub 2019 Jan 6. PMID 30625297